CLINICAL TRIAL: NCT02589314
Title: Effect of Mechanical Periodontal Therapy in the Microbiological, Immunocellular and Immunoglobulin Profiles and in the Dosage of Pro and Anti-inflammatory Cytokines From Peripheral Blood and Saliva of Subjects With Chronic Periodontitis and Diabetes Type 2
Brief Title: Effect of Periodontal Therapy in the Systemic Status of Individuals With Chronic Periodontitis and Diabetes Type 2
Status: Terminated | Type: Observational
Why Stopped: We could not achieve the number of participants necessary to continue with the study and limited money to continue with the study
Sponsor: University of Brasilia (Other)
Collaborators: Catholic University of Brasília (Other); Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Priscilla Farias Naiff, PhD student, University of Brasilia
Other Study IDs: CAAE 46609515.7.0000.0030
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Chronic Periodontitis; Diabetes Type 2
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2

GROUPS / COHORTS (1):
- root planning
  Interventions: Device: Mechanical periodontal therapy; Procedure: nonsurgical periodontal therapy

INTERVENTIONS:
Device: Mechanical periodontal therapy
  Other Names: periodontal debridment
Procedure: nonsurgical periodontal therapy

SUMMARY:
This study will evaluate if periodontal mechanical treatment is capable to alter immunological and genetical parameters related to systemic health in patients with chronic periodontitis ant diabetes type 2.

ELIGIBILITY:
Inclusion Criteria:

Periodontitis group:

* Minimum of 15 teeh;
* At least 30% of sites with periodontal probing depth ≥ 4 mm and at least two teeth with CAL ≥ 3 mm; Age ≥30 years;

Control group:

* Systemically healthy;
* 20 teeth;
* Probing depth ≤3 mm, clinical attachment level ≤3 mm , ≤10% of sites with bleeding on probing.

Exclusion Criteria:

* Periodontal treatment in the last six months;
* Continued use of medications such as antibiotics, immunomodulatory, anti-inflammatory drugs or corticosteroids in the last three months;
* Systemic diseases that interfere with periodontal condition, except for diabetes for the test group (HIV, cancer, immune disorders, acute infections, severe allergies, gastrointestinal or kidney disease, morbid obesity [BMI 40 kg / m2] or underweight [evil nourished BMI <18.5 kg / m2], etc.); Pregnant or lactating; smoking; Age <30 years; Indigenous groups.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Evidence of alteration in periodontal pathogens by PCR | One year
  Evaluate wich periodontal pathogens are detected before and after treatment
Evidence of alteration of immunocellular response by flowcytometry | one year
  Fenotype Monocytes, PMN, NK cells, T cells, B cells before and after periodontal treatment
Evidence of alteration on pro and anti-inflammatory cytokines by CBA | One year
  Dosage of cytokines before and after periodontal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Priscilla Farias Naiff, Brasília, Federal District, Brazil